CLINICAL TRIAL: NCT05734742
Title: Ttitudes Toward Obstructive Sleep Apnea-Related Cause of Road Traffic Accidents in Thailand Through Well Prepared Educational Video
Brief Title: Attitudes Toward Obstructive Sleep Apnea-Related Cause of Road Traffic Accidents in Thailand Through Well Prepared Educational Video
Acronym: AOSARTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Sarocha Vivatvakin, MD, Sarocha Vivatvakin, MD, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 796/65
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: OSA
Keywords: Attitudes; Obstructive sleep apnea (OSA); Survey; Traffic accident; Video
MeSH Terms: conditions — Behavior; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video (Experimental)
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — There were two videos including the first video "Sleep apnea Syndrome Driving Safety Picture Scroll" and the second video "Sleep apnea Syndrome and Traffic Accidents". The first video was approximately 3 minutes long. This video was suitable for all ages. It was an easy-to-understand video explaining the characteristics of OSA and its relationship with traffic accidents. The second video was the detailed video, which is approximately 20 minutes in duration. This video was suitable for those who desire to learn more about OSA. It can be used in various educational settings, including internal training and traffic safety workshops. Participants must watch at least the first video.

SUMMARY:
The goal of this descriptive, cross-sectional survey design is to determine the effect of public awareness video on the basic knowledge regarding sleep apnea syndrome or glaucoma and traffic accidents in normal population

The main questions it aims to answer are:

* To assess the attitudes toward the health-related cause of traffic accidents, mainly focused on obstructive sleep apnea and glaucoma among Thai people who viewed the local language translated versions of the public awareness video.
* To assess the feedbacks of the public awareness video.

Participants will be ask to complete a set of questionnaires containing 3 parts

* pre-test part
* educational video part
* post-test part

DETAILED DESCRIPTION:
Participants were asked to complete a set of questionnaires on obstructive sleep apnea and traffic accidents. The questionnaires were the modified version of the International Association of Traffic and Safety Sciences (IATSS) questionnaires. The questionnaires were designed as a self-administered questionnaire to access the attitudes and awareness of the health-related cause of traffic accidents focusing primarily on OSA. The questionnaire set was performed as an online questionnaire using Google Form. The questionnaires and videos were promoted through electronic posters. Participants were able to evaluate the questionnaire using the QR codes or links provided.

The questionnaire set consisted of three parts: 1) pre-test part (questionnaire before video watching), 2) educational video part (consisting of two videos), and 3) post-test part (questionnaire after video watching).

Participants were asked to complete the pre-test questionnaire part, which contained 13 items including 6 items on demographics of participants (gender, age, home town, frequency of motor vehicle use, education level, and occupation), 1 item on the underlying diseases of OSA, 1 item testing basic knowledge about common OSA symptoms, and 5 items regarding attitudes about OSA before watching educational videos.

Upon completion of the pre-test questionnaires and before starting the post-test questionnaires, participants were directed to the educational videos which were embedded in the same google form after the pre-test questionnaire. The purpose of the videos was to provide basic knowledge and to raise awareness of the OSA-related cause of traffic accidents. There were two videos including the first video "Sleep apnea Syndrome Driving Safety Picture Scroll" and the second video "Sleep apnea Syndrome and Traffic Accidents". The first video was approximately 3 minutes long. This video was suitable for all ages. It was an easy-to-understand video explaining the characteristics of OSA and its relationship with traffic accidents. The second video was the detailed video, which is approximately 20 minutes in duration. This video was suitable for those who desire to learn more about OSA. It can be used in various educational settings, including internal training and traffic safety workshops. Participants must watch at least the first video.

After viewing the videos, the participants were directed to the post-test questionnaires in the same google form. The post-test questionnaires contained 22 items including 10 items on attitudes about OSA or glaucoma (containing 5 same items as the pre-test questionnaires) and 12 items on video feedback. In conclusion, this questionnaire set consisted of 33 questions.

ELIGIBILITY:
Inclusion Criteria:

* employees of King Chulalongkorn Memorial Hospital
* aged ≥ 18 years

Exclusion Criteria:

* unable to cooperate to answer the questionnaires
* unable to view the videos

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
attitudes | one day
  attitudes toward the health-related cause of traffic accidents, mainly focused on OSA among Thai people who viewed these public awareness videos

SECONDARY OUTCOMES:
video feedback | one day
  feedback of the public awareness videos

CONTACTS AND LOCATIONS:
Overall Officials: Sarocha Vivatvakin, Principal Investigator — Department of Medicine, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No